CLINICAL TRIAL: NCT05247749
Title: Clinical Investigation to Evaluate the CONVIVO System for Discrimination of Normal Tissues From Abnormal Tissues During Brain Tumor Resection
Brief Title: CONVIVO System to Discriminate Healthy Tissues vs Tumor Tissues During Brain Tumor Resection
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Regulatory
Sponsor: Stanford University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB-48092; BRN0044 (Other: OnCore); IRB-48092 (Other: Stanford IRB)
Record Dates: First submitted 2022-02-09; First posted 2022-02-21 (Actual); Last update posted 2022-02-21 (Actual); Status verified 2022-02

CONDITIONS: Brain Tumor
MeSH Terms: conditions — Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Convivo Imaging (Experimental): The brain area that the operating surgeon plans to resect will be scanned using the CONVIVO device
  Interventions: Device: CONVIVO Confocal Endomicroscopy System

INTERVENTIONS:
Device: CONVIVO Confocal Endomicroscopy System — Confocal Laser Endomicroscopy (CEM) system intended for viewing intra-operative blood flow in the cerebral vascular area. Manufacturer - Zeiss

SUMMARY:
The purpose of the study is to do a direct comparison of the CONVIVO system (camera imaging device) with our normal Stanford pathology process. CONVIVO system is being tested to see if the device creates the images very quickly by touching a special camera to the surgical wound.

DETAILED DESCRIPTION:
Primary Objective:

The primary objective of this study is to determine the feasibility of using the CONVIVO imaging system to identify tumor type.

Secondary Objective: The secondary objectives are to determine the average time needed for tissue visualization with the CONVIVO system as compared to standard cryosectioning, and to describe the ability of the CONVIVO imaging

-To describe the ability of the CONVIVO imaging system to generate readable images.

ELIGIBILITY:
Inclusion Criteria:

* The subject demonstrates the ability to understand and the willingness to sign a written informed consent document.
* The subject is suspected to be suffering from following brain tumor: low-grade glioma, high grade-glioma, metastases, or meningioma.
* The subject has been deemed eligible for surgical resection by a practicing Stanford physician.
* Macroscopic tumor visualization using IV infusion of 500mg sodium fluorescein is planned as part of the subject's standard of care treatment.
* The subject is older than 18 years.
* The subject is receiving their surgery at Stanford Hospital.

Exclusion Criteria:

* Patients with any kind of contraindication to the use of fluorescein

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-05 (Estimated); Primary Completion 2022-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
Feasibility of using the CONVIVO imaging system to identify tumor tissue identified by the operating surgeon | 12 months
  Feasibility is defined as a match between the pathologist determination of a mock diagnosis of type of tumor using CONVIVO images of the planned resection area and the pathologist's cryosection-derived diagnosis used in the course of surgery. This outcome will be expressed as a number without dispersion.

SECONDARY OUTCOMES:
Average time needed for tissue visualization with the CONVIVO system as compared to standard cryosectioning | 12 months
  Time for tissue visualization with CONVIVO system: defined as the total number of minutes from start of imaging device use to mock diagnosis. This is calculated by summing the number of minutes from the start of imaging device use to the end of imaging device use in the operating room and the number of minutes from the neuropathologist's start of image review to arrival at a mock diagnosis.
  Time for standard cryosectioning: defined as the total number of minutes required for standard cryosectioning. This is calculated by summing the number of minutes from when the operating surgeon contacts the neuropathology department to request a frozen section analysis of tissue and ends when the neuropathology department calls the operating room with a suspected diagnosis, as measured by study personnel present in the operating room during the surgery
Ability of the CONVIVO system capture a readable image | 12 months
  A readable image is defined as an image from which a neuropathologist can make a mock diagnosis. This will be reported as a number without dispersion.

CONTACTS AND LOCATIONS:
Overall Officials: Gordon Li, Principal Investigator — Stanford Universiy

IPD SHARING:
Plan to Share IPD: No